CLINICAL TRIAL: NCT06353243
Title: Pilot of the Bilateral Infant Stimulation Study (BLISS): A Parent Provided Positive-Touch Intervention Targeting Stress in the Neonatal Intensive Care Unity (NICU)
Brief Title: Bilateral Infant Stimulation Study
Acronym: BLISS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kristen Mackiewicz Seghete, Principle Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00022901
Record Dates: First submitted 2024-03-28; First posted 2024-04-09 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Parent-Child Relations; Preterm Birth; Stress Reaction; Hospitalism in Children
Keywords: neonates; heart rate variability; bilateral stimulation; positive touch; NICU
MeSH Terms: conditions — Premature Birth; Fractures, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bilateral alternating Stimulation (Experimental): positive touch intervention provided by parent to infant using alternating stimulation
  Interventions: Behavioral: Bilateral alternating stimulation

INTERVENTIONS:
Behavioral: Bilateral alternating stimulation — positive touch intervention provided by parent to infant using alternating stimulation

SUMMARY:
This study will investigate stress that parents of children admitted to the neonatal intensive care unit (NICU) experience. Investigation of a novel intervention of using bilateral alternating stimulation to reduce parental stress and anxiety and increase bonding/attachment in NICU. Evaluate parental stress and feelings of bonding using surveys before and after the intervention. Intervention will be done at neonate's bedside while admitted to the NICU. Vital sign data will be collected as a marker of parent and neonate's stress response during the intervention.

DETAILED DESCRIPTION:
Objectives:

1. Examine the effect of a bilateral alternating stimulation (BAS) NICU intervention on parental anxiety and psychological distress in the NICU using biological and self-report measurements.
2. Examine the effect of a bilateral alternating stimulation NICU intervention on infants' physiological stress response after parental engagement in the BAS intervention with the infant.

This is a pilot study of bilateral alternating stimulation (BAS) examining the effectiveness as a therapeutic intervention for parental and infant stress in the NICU. It is a single arm design. Participants include parents and their infant that is currently admitted to the NICU. All participants will engage in parent-neonate intervention session, following this, infants will complete a delayed comparison arm (control session) with the interventionist. Infants currently admitted to NICU will be screened for eligibility, and if eligible, the families will be approached for enrollment. Families that enroll will be scheduled for one study session. During study session, parents will wear a heart rate monitor, complete psychologic scales of anxiety, stress, and feelings of closeness to thier infant, parents will be trained on the intervention and then engage in the intervention with their infant. Continuous vital signs will be collected for infant throughout the study session. After the intervention, parents will complete psychologic scales and satisfaction scales. Infants will then be scheduled for follow-up session where an interventionist will engage infant in intervention and vital signs will be collected throughout.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the NICU at the time of study
* greater than 34 weeks gestational age and less than 43 weeks gestational age
* within 4 weeks of admission to NICU at time of initial contact
* have parent or legal guardian willing and able to participate in the study

Exclusion Criteria:

* those who are less than 3 days postop from surgical procedures
* current use of psychotropic medications or medications that affect the central nervous system (CNS)
* CNS anomaly.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Parental anxiety | Administered immediately prior to engagement in study intervention activities and within 2 minutes post intervention
  Visual Analog Scale- Anxiety (VAS-A). The VAS scale asks participants to rate current anxiety on a horizontal line ranging from "calm" and "anxious" with scores between 0-100, with higher scores indicating higher levels of anxiety.
Physiologic stress response | total length of recording approximately 20 minutes for each participate, analysis will look at several minute epochs prior to and following intervention
  heart rate variability variable- the root mean square of successive diﬀerences (RMSSD) which reﬂects vagal tone
Parental distress | Administered immediately prior to engagement in study intervention activities and within 2 minutes post intervention
  Distress Thermometer

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health and Science University Neonatal Intensive Care Unit, Portland, Oregon, United States